CLINICAL TRIAL: NCT02572024
Title: The Effect of BATon BP and Sympathetic Function in Resistant Hypertension (The Nordic BAT Study)
Acronym: BAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Odense University Hospital (Other); University of Oslo (Other); University of Helsinki (Other); Sahlgrenska University Hospital (Other); Skane University Hospital (Other)
Responsible Party: Principal Investigator, Daniel Gordin, MD DMSc, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BATstudy
Record Dates: First submitted 2015-10-07; First posted 2015-10-08 (Estimated); Last update posted 2023-03-02 (Actual); Status verified 2022-03

CONDITIONS: Resistant Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Baroreflex activation therapy (Active Comparator): BAT ON
  Interventions: Device: BAT
- Placebo (Placebo Comparator): BAT OFF
  Interventions: Other: Placebo

INTERVENTIONS:
Device: BAT — Baroreflex activation therapy device ON
  Arms: Baroreflex activation therapy
Other: Placebo — Baroreflex activation therapy device OFF
  Arms: Placebo

SUMMARY:
Resistant hypertension (RH) affects some 10% to 15% of all patients with hypertension. These patients are at a clearly increased risk for end organ damage and mortality. Furthermore, arterial hypertension is a multifactorial disease including genetic, lifestyle, dietary, metabolic, and sympathetic factors. However, the current treatment modalities have not been optimal in targeting the compensatory changes in sympathetic nervous system function and new strategies have been warranted.

Baroreflex activation therapy (BAT) is a special treatment option for some patients with RH that modulates the autonomic nervous system to restore sympathovagal balance. Notably, in BAT both long-term safety and efficacy in a large-scale, randomized, double blind, controlled trial has been shown. However, the trial design and BAT methodology resulted in that the first generation Rheos® system did not achieve the prespecified endpoints for short-term safety and efficacy.

Notably, a second-generation minimally invasive BAT system (Barostim Neo®) has now been developed to address these limitations although randomized, double blind, controlled clinical trials are still lacking. Noteworthy, in the recent European Society of Hypertension/European Society of Cardiology (ESH/ESC) Guidelines for the management of arterial hypertension, carotid baroreceptor stimulation is mentioned as one of the options to treat resistant hypertension.

Based on these data the aim of this randomized, double-blind, parallel-design clinical trial is to examine the effect of BAT compared to continuous pharmacotherapy on blood pressure, as well as arterial and cardiac function and structure using non-invasive high technology methodology, in a Nordic multicentre study.

This study will include 100 patients with RH (20 from Helsinki). Eligible patients are between 18 and 70 years and have a daytime systolic ambulatory blood pressure 145 mmHg or more, and/or a daytime diastolic ambulatory blood pressure of 95 mmHg or more, after witnessed intake of antihypertensive treatment (including at least 3 antihypertensive drugs preferably including a diuretic), with no changes in medication for a minimum of 4 weeks prior to enrolment. Patients with severe renal insufficiency, type 1 diabetes, psychiatric illness, severe cardiovascular disease, or any complication that is a risk to the planned surgery are exclusion criteria.

The primary end point is to test whether BAT reduces 24-hour systolic ambulatory blood pressure at 8 months of follow-up compared to continuous pharmacotherapy. Secondary end points are to test whether BAT reduces home blood pressure during follow-up compared to continuous pharmacotherapy, whether BAT reduces office blood pressure during follow-up compared to continuous pharmacotherapy, and the effect of BAT on autonomic function measured as eg. baroreflex sensitivity and heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients have a daytime systolic ambulatory blood pressure 145 mmHg or more, and/or a daytime diastolic ambulatory blood pressure of 95 mmHg or more, after witnessed intake of antihypertensive treatment (including at least 3 antihypertensive drugs preferably including a diuretic), with no changes in medication for a minimum of 4 weeks prior to enrolment.

Exclusion Criteria:

* Patients with secondary causes of hypertension will be excluded.
* Further exclusion criteria are renal insufficiency with an estimated glomerular filtration rate ≤30 ml/min/1.73 m2 (using the Chronic Kidney Disease Epidemiology [CKD-EPI] formula), untreated sleep apnoea, pregnancy, type 1 diabetes, alcohol or substance abuse or psychiatric illnesses, other heart rhythm than sinus (well controlled atrial fibrillation is not a contraindication), uncontrolled systolic heart failure (or an ejection fraction of less than 40% in echocardiography), aortic stenosis (mean gradient more than 25 mmHg in echocardiography).
* Myocardial infarction, hypertensive crisis, symptomatic orthostatic hypotension, unstable angina, syncope, or cerebral vascular accident within the 3 months before enrolment will also be exclusion criteria.
* Furthermore, known or suspected baroreflex failure or autonomic neuropathy, carotid artery stenosis as well as prior surgery, radiation, or endovascular stent placement in the carotid sinus region on both sides, as well as any complication that is a risk to the planned surgery are exclusion criteria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2022-11 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
Change in systolic ambulatory blood pressure in response to BAT therapy | 8 months
  Unit: mmHg

SECONDARY OUTCOMES:
Change in systolic ambulatory blood pressure in response to BAT therapy | 19 months
  Unit: mmHg
Change in home/office blood pressure in response to BAT therapy | 19 months
  Unit: mmHg
Change in autonomic function in response to BAT therapy | 19 months
  Unit: ms/mmHg

CONTACTS AND LOCATIONS:
Locations (5):
- Odense University Hospital, Odense, Denmark
- Helsinki University Central Hospital, Helsinki, Finland
- University of Oslo, Oslo, Norway
- Sweden (2):
  - Sahlgrenska University Hospital, Sweden, Gothenburg
  - Skåne University Hospital, Malmo